CLINICAL TRIAL: NCT02362412
Title: Study of FK949E - An Open-label, Two-way Crossover Study to Evaluate the Effects of Switching Different Strength Forms of FK949E in Bipolar Disorder Patients With Major Depressive Episodes
Brief Title: Study to Evaluate the Effects of Switching Different Strength Forms of FK949E in Bipolar Disorder Patients With Major Depressive Episodes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6949-CL-0023
Record Dates: First submitted 2015-02-03; First posted 2015-02-12 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Bipolar Depression
Keywords: major depressive episodes; FK949E; quetiapine; bipolar depression; bipolar disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FK949E 50 MG / FK949E 150 MG (Experimental): Participants who received the 50 mg tablet once daily during Treatment Period II (8 weeks) and 150 mg tablet once daily during Treatment Period III (8 weeks).
  Interventions: Drug: FK949E
- FK949E 150 MG / FK949E 50 MG (Experimental): Participants who received the 150 mg tablet once daily during Treatment Period II (8 weeks) and 50 mg tablet once daily during Treatment Period III (8 weeks).
  Interventions: Drug: FK949E

INTERVENTIONS:
Drug: FK949E — A tablet containing 50 mg or 150 mg of quetiapine taken orally.
  Other Names: quetiapine

SUMMARY:
The purpose of this study was to evaluate the efficacy, safety, and pharmacokinetics of switching FK949E (sustained-release quetiapine) 50-mg and 150-mg tablets to the other tablet at the equivalent total daily dose in bipolar disorder patients with major depressive episodes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar I or II disorder as specified in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR), with a major depressive episode.
* Able to participate in the study with understanding of and compliance with subject requirements during the study in the investigator's or subinvestigator's opinion.

Exclusion Criteria:

* Concurrent or previous history of DSM-IV-TR Axis I disorders, except bipolar disorder, within the last 6 months before informed consent.
* Concurrence of DSM-IV-TR Axis II disorder that is considered to greatly affect patient's current mental status.
* The Young Mania Rating Scale (YMRS) total score of 13 points or more.
* Nine or more mood episodes within the last 12 months before informed consent.
* Lack of response to at least 6-week treatment with at least 2 antidepressants for the current major depressive episode in the investigator's or subinvestigator's opinion.
* The current major depressive episode persisting for less than 4 weeks before informed consent.
* History of substance dependence (other than caffeine and nicotine) or alcohol abuse or dependence.
* Treatment with a depot antipsychotic within the last 49 days before the start of the pre-treatment observation period.
* Unable to suspend antipsychotics or antidepressants after the start of the pre-treatment observation period.
* Treatment with more than one of the following three drugs, mood stabilizers (lithium carbonate and/or sodium valproate) and lamotrigine, if these drugs, except one of either drugs, cannot be suspended after the start of the pre-treatment observation period.
* Unable to suspend antiepileptics (except lamotrigine and sodium valproate), antianxiety agents, hypnotics, sedatives, psychostimulants, antiparkinsonian agents, cerebral ameliorators, antidementia agents, or anorectics, except those specified as conditionally-allowed concomitant drugs, from 7 days before the start of the pre-treatment observation period.
* Unable to suspend CYP3A4 inhibitors or inducers, or monoamine oxidase (MAO) inhibitors from 7 days before the start of the pre-treatment observation period.
* Electroconvulsive therapy within the last 83 days before the start of the pre-treatment observation period.
* A possible need of psychotherapy during the study period (unless the therapy has been commenced at least 83 days before the start of the pre-treatment observation period).
* The Hamilton Depression Rating Scale (HAM-D17) suicide score of 3 points or more, history of suicide attempt within the last 6 months before informed consent, or the risk of suicide in the investigator's or subinvestigator's opinion.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2016-02-06 (Actual); Study Completion 2016-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Fukushima
  - Kanagawa
  - Kumamoto
  - Kyoto
  - Osaka
  - Tokushima
  - Tokyo

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Fukushi R, Nomura Y, Katashima M, Komatsu K, Sato Y, Takada A. Approach to Evaluating QT Prolongation of Quetiapine Fumarate in Late Stage of Clinical Development Using Concentration-QTc Modeling and Simulation in Japanese Patients With Bipolar Disorder. Clin Ther. 2020 Aug;42(8):1483-1493.e1. doi: 10.1016/j.clinthera.2020.06.002. Epub 2020 Aug 11. PMID 32792252
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with documented clinical diagnosis meeting the DSM-IV-TR criteria for bipolar I disorder or bipolar II disorder, with most recent episode depressed (296.50 to 296.54 or 296.89) confirmed by the Mini-International Neuropsychiatric Interview (M.I.N.I.) were recruited from 10 sites in Japan.
Pre-assignment Details: After informed consent was obtained and prior to randomization in Treatment Period II, participants entered Treatment Period I (4 weeks) to allow a dose titration and reduction for adjusting the dosage regimen of FK949E. Two participants did not enter Treatment Period II (due to an adverse event and withdrawal of consent, respectively).
Period: Treatment Period II
Arm/Group | FK949E 50 mg / FK949E 150 mg | FK949E 150 mg / FK949E 50 mg
Started | 9 | 11
TREATED | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0
Period: Treatment Period III
Arm/Group | FK949E 50 mg / FK949E 150 mg | FK949E 150 mg / FK949E 50 mg
Started | 9 | 11
TREATED | 9 | 11
Completed | 9 | 10
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who received either FK949E 50 mg tablets or FK949E 150 mg tablets once daily. The analysis population was the Full Analysis Set (FAS), which consisted of all participants who received at least one dose of the study drug and who had at least one efficacy measurement after the start of treatment with the study drug.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
MONTGOMERY-ASBERG DEPRESSION RATING SCALE (MADRS) TOTAL SCORE [Mean (Standard Deviation); unit: UNITS ON A SCALE] — The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms
  UNITS ON A SCALE | 19.8 (8.6)
HAMILTON DEPRESSION SCALE (HAM-D17) TOTAL SCORE [Mean (Standard Deviation); unit: UNITS ON A SCALE] — The HAM-D17 is a clinician-rated 17-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52 with lower scores indicating less depressive symptoms.
  UNITS ON A SCALE | 14.5 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms.
Time Frame: Week 8 of each treatment period (Week 12 and Week 20)
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (95% Confidence Interval); unit: UNITS ON A SCALE
Groups:
- FK949E 50 mg Tablets: Participants who received FK949E 50 mg tablets once daily in either Treatment Period II (8 weeks) or Treatment Period III (8 weeks).
- FK949E 150 mg Tablets: Participants who received FK949E 150 mg tablets once daily in either Treatment Period II (8 weeks) or Treatment Period III (8 weeks).
Arm/Group | FK949E 50 mg Tablets | FK949E 150 mg Tablets
Number analyzed (Participants) | 20 | 20
UNITS ON A SCALE | 7.4 [4.4 to 10.4] | 7.9 [5.0 to 10.9]
Statistical Analysis 1: Comparison: FK949E 50 mg Tablets vs FK949E 150 mg Tablets; Test type: Superiority or Other; p-value was not adjusted; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-3.4 to 2.3] — Analysis of variance with treatment sequence, time point, and formulation as fixed effects and patient as a random effect using the data at Week 12 and Week 20 of the treatment period

2. Secondary Outcome: Hamilton Depression Scale (HAM-D17)
Description: The HAM-D17 is a clinician-rated 17-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52 with lower scores indicating less depressive symptoms.
Time Frame: Week 8 of each treatment period (Week 12 and Week 20)
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | FK949E 50 mg Tablets | FK949E 150 mg Tablets
Number analyzed (Participants) | 20 | 20
Units on a scale | 5.5 [3.4 to 7.5] | 5.4 [3.4 to 7.3]
Statistical Analysis 1: Comparison: FK949E 50 mg Tablets vs FK949E 150 mg Tablets; Test type: Superiority or Other; Least Squares Mean Difference = 0.1, 95% CI 2-sided [-1.7 to 1.9] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Clinical Global Impression-Bipolar-Severity of Illness (CGI-BP-S): Overall Bipolar Illness
Description: The CGI-BP-S is a scale which assesses a participant's severity of their overall bipolar illness, depression, and mania as assessed by the clinician using a scale from with the scale from 1 (Normal, not ill) to 7 (very severely ill).
Time Frame: Week 8 of each treatment period (Week 12 and Week 20)
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | FK949E 50 mg Tablets | FK949E 150 mg Tablets
Number analyzed (Participants) | 20 | 20
Units on a scale | 2.1 [1.7 to 2.5] | 2.0 [1.7 to 2.4]
Statistical Analysis 1: Comparison: FK949E 50 mg Tablets vs FK949E 150 mg Tablets; Test type: Superiority or Other; Least Squares Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.4] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Clinical Global Impression-Bipolar-Severity of Illness (CGI-BP-S):Depression
Description: as for outcome 3
Time Frame: Week 8 of each treatment period (Week 12 and Week 20)
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | FK949E 50 mg Tablets | FK949E 150 mg Tablets
Number analyzed (Participants) | 20 | 20
Units on a scale | 2.1 [1.7 to 2.5] | 2.0 [1.7 to 2.4]
Statistical Analysis 1: Comparison: FK949E 50 mg Tablets vs FK949E 150 mg Tablets; Test type: Superiority or Other; Least Squares Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.4] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Clinical Global Impression-Bipolar-Severity of Illness (CGI-BP-S): Mania
Description: as for outcome 3
Time Frame: Week 8 of each treatment period (Week 12 and Week 20)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FK949E 50 mg Tablets | FK949E 150 mg Tablets
Number analyzed (Participants) | 20 | 20
Units on a scale | 1.0 (0.0) | 1.0 (0.0)

6. Secondary Outcome: Clinical Global Impression-Bipolar-Change (CGI-BP-C):Overall Bipolar Illness
Description: The CGI-BP-C is a scale which assesses the degree of change or improvement from baseline for each of overall bipolar illness, depression and mania, by grading it using 8 grades, from 1 (very much improved) to 7 (very much worse) or 8 (not applicable). Grade 8 (not applicable) was regarded as a missing value for purposes of calculating the mean score.
Time Frame: Week 8 of each treatment period (Week 12 and Week 20)
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | FK949E 50 mg Tablets | FK949E 150 mg Tablets
Number analyzed (Participants) | 20 | 20
Units on a scale | 2.0 [1.6 to 2.5] | 2.0 [1.6 to 2.5]
Statistical Analysis 1: Comparison: FK949E 50 mg Tablets vs FK949E 150 mg Tablets; Test type: Superiority or Other; Least Squares Mean Difference = -0.0, 95% CI 2-sided [-0.5 to 0.5] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Clinical Global Impression-Bipolar-Change (CGI-BP-C):Depression
Description: as for outcome 6
Time Frame: Week 8 of each treatment period (Week 12 and Week 20)
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | FK949E 50 mg Tablets | FK949E 150 mg Tablets
Number analyzed (Participants) | 20 | 20
Units on a scale | 2.0 [1.6 to 2.5] | 2.0 [1.6 to 2.5]
Statistical Analysis 1: Comparison: FK949E 50 mg Tablets vs FK949E 150 mg Tablets; Test type: Superiority or Other; Least Squares Mean Difference = -0.0, 95% CI 2-sided [-0.5 to 0.5] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Clinical Global Impression-Bipolar-Change (CGI-BP-C):Mania
Description: as for outcome 6
Time Frame: Week 8 of each treatment period (Week 12 and Week 20)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FK949E 50 mg Tablets | FK949E 150 mg Tablets
Number analyzed (Participants) | 20 | 20
Units on a scale | 4.0 (0.0) | 4.0 (0.0)

9. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any undesirable or unintended sign (including abnonmal laboratory test values), symptom, or disease occurring while the study drug was administered, regardless of whether or not there was a causal relationship with the study drug. A serious AE is defined as a an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, was life-threatening, required or prolonged hospitalization or was considered medically important.
Time Frame: Up to 22 weeks
Population: Safety Analysis Set (SAF), which included participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- Treatment Period II FK949E 50 mg: Participants who received FK949E 50 mg tablets once daily during Treatment Period II (8 weeks).
- Treatment Period II FK949E 150 mg: Participants who received FK949E 150 mg tablets once daily during Treatment Period II (8 weeks).
- Treatment Period III FK949E 150 mg: Participants who received FK949E 150 mg tablets once daily during Treatment Period III (8 weeks).
- Treatment Period III FK949E 50 mg: Participants who received FK949E 50 mg tablets once daily during Treatment Period III (8 weeks).
Arm/Group | Treatment Period II FK949E 50 mg | Treatment Period II FK949E 150 mg | Treatment Period III FK949E 150 mg | Treatment Period III FK949E 50 mg
Number analyzed (Participants) | 9 | 11 | 9 | 11
Participants
  Any AE | 1 | 2 | 5 | 2
  Drug-related AEs | 0 | 1 | 2 | 0
  Deaths | 0 | 0 | 0 | 0
  Serious AEs | 0 | 0 | 0 | 0
  Drug-related SAEs | 0 | 0 | 0 | 0
  AEs that caused study drug discontinuation | 0 | 0 | 0 | 0
  Drug-related AEs that caused study drug discont. | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 7 days after last dose of study drug (22 weeks)
Groups:
- Treatment Period II FK949E 150 mg: Participants who received FK949E 150 mg tablets once daily duringr Treatment Period II (8 weeks).
Arm/Group | Treatment Period II FK949E 50 mg | Treatment Period II FK949E 150 mg | Treatment Period III FK949E 150 mg | Treatment Period III FK949E 50 mg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 1/9 | 2/11 | 5/9 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period II FK949E 50 mg (N=9) | Treatment Period II FK949E 150 mg (N=11) | Treatment Period III FK949E 150 mg (N=9) | Treatment Period III FK949E 50 mg (N=11)
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment.